CLINICAL TRIAL: NCT00891033
Title: Phase I Exploratory Study of Panobinostat IV in Combination With Bortezomib in Relapsed/Refractory Multiple Myeloma Patients
Brief Title: Panobinostat/Velcade in Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated because the drug company stopped making the study drug
Sponsor: University of Arkansas (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI32829
Record Dates: First submitted 2009-04-28; First posted 2009-04-30 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Multiple Myeloma
Keywords: cancer
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — Bortezomib; Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): 1 mg/m2 IV Bortezomib on days 1, 4, 8, and 11 of Cycles 1 and 2 and 5 mg/m2 IV Panobinostat on days 1 and 8 of Cycle 2.
  Interventions: Drug: Bortezomib (Velcade); Drug: Panobinostat
- Cohort 2 (Experimental): 1 mg/m2 IV Bortezomib on days 1, 4, 8, and 11 of Cycles 1 and 2 and 10 mg/m2 IV Panobinostat on days 1 and 8 of Cycle 2.
  Interventions: Drug: Bortezomib (Velcade); Drug: Panobinostat
- Cohort 3 (Experimental): 1 mg/m2 IV Bortezomib on days 1, 4, 8, and 11 of Cycles 1 and 2 and 15 mg/m2 IV Panobinostat on days 1 and 8 of Cycle 2.
  Interventions: Drug: Bortezomib (Velcade); Drug: Panobinostat
- Cohort 4 (Experimental): 1 mg/m2 IV Bortezomib on days 1, 4, 8, and 11 of Cycles 1 and 2 and 20 mg/m2 IV Panobinostat on days 1 and 8 of Cycle 2.
  Interventions: Drug: Bortezomib (Velcade); Drug: Panobinostat

INTERVENTIONS:
Drug: Bortezomib (Velcade) — During the study Bortezomib will be administered intravenously as a 3-5 second bolus IV injection, at a dose of 1.0 mg/m2 on days 1, 4, 8, and 11 of each 21-day treatment cycle.
  Other Names: Velcade
Drug: Panobinostat — During the study, panobinostat IV will be administered intravenously as once daily on (day 1 and 8 of the 21 day cycle 2 and beyond). Patients enrolled on first group will receive 5 mg/m2 panobinostat IV, second group 10 mg/m2 panobinostat IV, third group 15 mg/m2 panobinostat IV and the fourth group 20 mg/m2 panobinostat IV. Each infusion of panobinostat will be administered over 30 minutes.

SUMMARY:
Multiple myeloma (MM) accounts for approximately 1% of all malignancies and 10% of hematological tumors, representing the second most frequently occurring hematological malignancy in the United States. At any one time, 50,000 people suffer from MM, and approximately 15,000 are diagnosed each year. The median age is approximately 65 years, although occasionally MM occurs in the second decade of life.

Bortezomib and panobinostat intravenous (IV) are active agents in multiple myeloma and appear to work through different biochemical pathways, suggesting that there may be a synergistic effect using the combination. Both compounds have shown anabolic bone effect, which has been associated to significant anti-myeloma activity.

Primary objectives:

* To assess the toxicity of bortezomib combined with one of 4 doses of panobinostat IV in patients with relapsed/refractory multiple myeloma, and
* To find the most appropriate doses of bortezomib and panobinostat IV in the combination.

Secondary objective:

* To assess the effect of bortezomib in combination with panobinostat IV on inducing osteoblast activation in patients with relapsed/refractory myeloma.

DETAILED DESCRIPTION:
The objective of this study is to identify the maximum tolerated dose (MTD) and assess the feasibility and toxicity experience for patients with refractory multiple myeloma treated with bortezomib and one of three doses of panobinostat IV.

Sample Size:

This study will accrue up to 24 patients, in 4 groups of up to 6 patients each, depending on experiences of DLT. Patients will be studied as follows, Group 1: Bortezomib 1.0 mg/m2 and panobinostat IV 5 mg/m2 IV, Group 2: Bortezomib 1.0 mg/m2and panobinostat IV 10 mg/m2 IV, Group 3: Bortezomib 1.0 mg/m2 and panobinostat IV 15 mg/m2 IV and Group 4: Bortezomib 1.0 mg/m2 and panobinostat IV 20 mg/m2 IV. Bortezomib will be given on days 1, 4, 8, and 11 during cycle 1 and cycle 2, and panobinostat will be given on days 1 and 8 of the second cycle.

If the MTD is not reached with the first group, the second group will be enrolled and will receive bortezomib1.0 mg/m2 with escalation of panobinostat IV as described above.

Patient population:

Patient's with relapsed/refractory multiple myeloma with at least one line of prior therapy.

Inclusion and exclusion criteria:

Patients must have baseline evaluations performed prior to the first dose of study drug and must meet all inclusion and exclusion criteria. Results of all baseline evaluations, which assure that all inclusion and exclusion criteria have been satisfied, must be reviewed by the principal investigator prior to enrollment of that patient. In addition, the patient must be thoroughly informed about all aspects of the study, including the study visit schedule and required evaluations and all regulatory requirements for informed consent. The written informed consent must be obtained from the patient prior to enrollment. The following criteria apply to all patients enrolled onto the study unless otherwise specified.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed/refractory multiple myeloma to at least one line of prior therapy
2. Male or female patients aged ≥ 18 years old
3. Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
4. Patients are allowed to receive growth factors (erythropoietin hormones, GCSF and GMCSF)
5. Patients must meet the following laboratory criteria:

   * ANC ≥ 1.5 x 109/L
   * Hemoglobin ≥ 9 g/dl
   * Platelets ≥ 100x 109/L
   * Calculated CrCl > 50 mL/min (MDRD Formula)
   * AST and ALT ≤ 2.5 x ULN
   * Serum bilirubin < 2.0 x ULN
   * Albumin > 3.0 g/dl
   * Serum potassium ≥ LLN for the institution
   * Total serum calcium [corrected for serum albumin] or ionized calcium ≥LLN, for the institution
   * Serum magnesium ≥ LLN for the institution
   * Serum phosphorus ≥ LLN for the institution
   * TSH ≤ LLN and free T4 within normal limits. Patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism
6. Baseline MUGA or ECHO must demonstrate LVEF ≥ the lower limit of the institutional normal
7. History of histologically documented MM with relapsed or progressive disease after at least one line of prior therapy
8. Patient has measurable disease in which to capture response, defined as one or more of the following:

   1. Serum M-protein level ≥ 0.5 gm/dl (10.0 g/L) measured by serum protein electrophoresis or immunoglobulin electrophoresis; or
   2. Urinary M-protein excretion ≥ 200 mg/24 hrs; or
   3. Bone marrow plasmacytosis of ≥ 30% by bone marrow aspirate and/or biopsy; or
   4. Serum Free Light Chains (By the Freelite test) > 2X ULN, in the absence of renal failure
9. Performance status of ≤ 2 as per ECOG scale, unless PS of 3-4 based solely on bone pain
10. Patients must have signed an IRB approved written informed consent form and demonstrate willingness to meet follow-up schedule and study procedure obligations

Exclusion Criteria:

1. Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer
2. Patients who have received Velcade within 2 months of enrollment
3. Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first panobinostat IV treatment
4. Peripheral neuropathy > grade 2.
5. Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

   * Patients with congenital long QT syndrome
   * History or presence of sustained ventricular tachyarrhythmia. (Patients with a history of atrial arrhythmia are eligible but should be discussed with Novartis prior to enrollment)
   * Any history of ventricular fibrillation or torsade de pointes
   * Bradycardia defined as HR< 50 bpm. Patients with pacemakers are eligible if HR ≥ 50 bpm.
   * Screening ECG with a QTc > 450 msec
   * Right bundle branch block + left anterior hemiblock (bifascicular block)
   * Patients with myocardial infarction or unstable angina ≤ 6 months prior to starting study drug
   * Other clinically significant heart disease (e.g., CHF NY Heart Association class III or IV , uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
6. Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes or active or uncontrolled infection) including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol
7. Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug
8. Concomitant use of CYP3A4 inhibitors (See Appendix 2)
9. Patients who have received targeted agents within 2 weeks or within 5 half-lives of the agent and active metabolites (which ever is longer) and who have not recovered from side effects of those therapies.
10. Patients who have received either immunotherapy (e.g. vaccines) within < 8 weeks; chemotherapy within < 4 weeks; or radiation therapy to > 30% of marrow-bearing bone within < 2 weeks prior to starting study treatment; or who have not yet recovered from side effects of such therapies.
11. Patients with an active bleeding tendency or is receiving any treatment with therapeutic doses of sodium warfarin (Coumadin®) or coumadin derivatives. Low doses of Coumadin® (e.g. ≤ 2.0 mg/day) to maintain line patency (if applicable) is allowed.
12. Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
13. Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not using an effective method of birth control. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months). Women of childbearing potential must have a negative serum pregnancy test within 24hrs of receiving the first dose of study medication.
14. Male patients whose sexual partners are WOCBP not using effective birth control
15. Patients with a prior malignancy with in the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix)
16. Patients with known positivity for human immunodeficiency virus (HIV) ) or hepatitis C; baseline testing for HIV and hepatitis C is not required
17. Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff.
18. No concomitant use of bisphosphonates is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Toxicity of bortezomib combined with one of 3 doses of panobinostat IV as measured by the occurrence of dose-limiting toxicity (DLT) | up to 42 days (two 21-day cycles)
  DLT is defined as at least 2 of 6 patients within a group experiencing greater than or equal to grade 3 non-hematologic toxicity or greater than or equal to grade 4 hematologic toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Mauizio Zangari, MD, Principal Investigator — University of Utah
Locations (1):
- Myeloma Institute for Research and Therapy University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States